CLINICAL TRIAL: NCT04825340
Title: To Explore a Bridging Index for the Effectiveness of the Clinical Trial With Nasal Spray Lyophilized Live Attenuated Influenza Vaccine
Brief Title: To Explore a Bridging Index for the Effectiveness of the Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F202110111
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Randomized
Keywords: Influenza Vaccine Nasal Spray

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study vaccine (Experimental): Nasal Spray Lyophilized Live Attenuated Influenza Vaccine
  Interventions: Biological: Nasal Spray Lyophilized Live Attenuated Influenza Vaccine
- Placebo (Placebo Comparator): commercial normal saline
  Interventions: Biological: Nasal Spray Lyophilized Live Attenuated Influenza Vaccine

INTERVENTIONS:
Biological: Nasal Spray Lyophilized Live Attenuated Influenza Vaccine — 0.2 ml/vial, 0.2ml/dose/per person

SUMMARY:
To explore a bridging index for the effectiveness of the clinical trial with Nasal Spray Lyophilized Live Attenuated Influenza Vaccine

DETAILED DESCRIPTION:
With a randomized, blind, parallel placebo-controlled design, to screen the susceptible individuals aged 3~59 years old whose titers of either of Hi antibody level of H1N1, H3N2 or B are not higher than 1:10 prior immunization , in which all persons are to be assigned into the two subgroups (aged 3~17 and 18~59 years old) with radio of 1:1, individually. All persons of each age subgroups are to be randomly assigned into the two groups (vaccine or placebo group) with th radio of 2:1 via intranasal injection of one dose of the study vaccine or placebo. The blood samples are to be collected prior immunisation and on the 21st day post immunisation, individually, the nasopharyngeal swab samples are also to be done prior immunisation and on the 10th day and 21st day post immunisation, individually, and the levels of serum HI antibody and mucous sIgA antibody are to be compared between the two groups, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. healthy volunteer aged 3~59 years old；
2. no vaccination with any influenza vaccine within the past year；
3. no catching any influenza or flu like symptoms （axillary temperature ≥ 38℃， accompanied by cough or sore throat ）；
4. influenza susceptible individual（any serum Hi antibody level of H1N1, H3N2 and B≦1:10）；
5. with informed consent obtained from the volunteer and / or guardian；
6. willing of volunteers and / or guardians to comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

1. Known allergy individual to any ingredient of this product, including egg protein, subsidiary material and/or gentamycin sulfate;
2. patients with acute disease, severe chronic disease, acute attack of chronic disease and/or fever (axillary temperature ≥ 37.3℃ on the day of immunisation);
3. pregnancy (enquire);
4. patients with Leigh syndrome treated with aspirin or aspirin containing drugs;
5. patients with immunodeficiency or receiving immunosuppressive therapy;
6. patients with uncontrolled epilepsy and other progressive nervous system diseases, with a history of Guillain Barre syndrome;
7. patients with rhinitis or other nasal abnormalities judged by clinicians that may affect vaccination or sample collection;
8. accept any immunoglobulin and / or any blood products within 3 months, or plan to use them during the study (until post immunization blood sample collection);
9. .taking anti influenza drugs in the past 48 hours;
10. .any situation that the researchers believe may affect the study.

Ages: 3 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-04-16 (Estimated); Primary Completion 2022-03-25 (Estimated); Study Completion 2022-03-25 (Estimated)

PRIMARY OUTCOMES:
The GMTs of serum HI antibodies of all H1N1, H3N2 and B | 0-21 days
  The GMTs of serum HI antibodies of all H1N1, H3N2 and B on the 21st day post immunization;
GMTs of HI sIgA antibodies of all H1N1, H3N2 and B | 10-21 days
  The mucous GMTs of HI sIgA antibodies of all H1N1, H3N2 and B on the 10th and 21st day post immunization;

SECONDARY OUTCOMES:
The ratios and 95% CI of the GMTs of serum HI antibodies of all H1N1, H3N2 and B | 0-21days
  The ratios and 95% CI of the GMTs of serum HI antibodies of all H1N1, H3N2 and B on the 21st day post immunization;